CLINICAL TRIAL: NCT05809180
Title: Prospective Exploratory Clinical Study of Orelabrutinib, Pomalidomide, Rituximab Combined With miniCHOP-like Regimen in Treatment-naive Elderly Patients With DLBCL
Brief Title: Pro-miniCHOP-like Regimen for Treatment-naive Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Jinzm 005
Record Dates: First submitted 2023-03-22; First posted 2023-04-12 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-02

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma; Orelabrutinib; pomalidomide; Rituximab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; orelabrutinib; pomalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rituximab(100mg), orelabrutinib(50mg), pomalidomide(4mg), miniCHOP-like (Experimental): 1. Phase I(induction therapy): Patients receive Rituximab on day 1, Pomalidomide on days 1-7 and oral administration of Orelabrutinib per day.
  2. Phase II(stratified response therapy):
     Part A: (25% or more reduction): Patients receive Pro-miniCHOP-like regimen every 21 days for 6 cycles.(Rituximab on day 1, Pomalidomide on days 1-7, Orelabrutinib per day till progression or intolerant toxicity, Cyclophosphamide on day 2, Doxorubicin/Doxorubicin Liposome on day 2, Vindesine on day 2 and Dexamethasone on days 2-6).
     Part B: (reduction less than 25%): Patients receive R-miniCHOP-like regimen every 21 days for 6 cycles.(Rituximab on day 1, Cyclophosphamide on day 2, Doxorubicin/Doxorubicin Liposome on day 2, Vindesine on day 2 and Dexamethasone on days 2-6).
  3. Phase III(maintenance and follow-up): Patients take Pomalidomide orally on days 1-7 in a cycle of 21 days for 2 years.
  Interventions: Drug: Rituximab; Drug: Orelabrutinib; Drug: Pomalidomide; Drug: Pro-miniCHOP-like regimen; Drug: R-miniCHOP-like regimen

INTERVENTIONS:
Drug: Rituximab — Rituximab 375mg/m2 ivgtt d1;
  Other Names: MabThera
Drug: Orelabrutinib — Orelabrutinib 150mg per day oral administration till progresses or intolerant toxicity;
  Other Names: Yinuokai
Drug: Pomalidomide — Pomalidomide 4mg d1-7 each cycle. After Phase II of treatment, single agent pomalidomide 4 mg d1-d7 in 21-day cycles for 2 years.
  Other Names: Anyve
Drug: Pro-miniCHOP-like regimen — rituximab 375mg/m2 ivgtt d1; orelabrutinib 150mg per day oral administration till progresses or intolerant toxicity; pomalidomide 4mg d1-7; cyclophosphamide 400mg/m2 ivgtt d2; doxorubicin 25mg/m2 ivgtt d2/ doxorubicin liposome 15 mg/m2 ivgtt d2; vindesine 2mg ivgtt d2; dexamethasone 10mg ivgtt d2-6.
Drug: R-miniCHOP-like regimen — rituximab 375mg/m2 ivgtt d1; cyclophosphamide 400mg/m2 ivgtt d2; doxorubicin 25mg/m2 ivgtt d2/ doxorubicin liposome 15 mg/m2 ivgtt d2; vindesine 2mg ivgtt d2; dexamethasone 10mg ivgtt d2-6.

SUMMARY:
The proposed study is a prospective, single-center and open-ended study in patients over the age of 70 with treatment-naive diffuse large B-cell lymphoma (DLBCL). This study intends to explore a new treatment pattern using Pro-miniCHOP-like regimen and simultaneously evaluate its safety and efficacy for future clinical practice.

DETAILED DESCRIPTION:
The study will start with an initial 21-days of induction therapy with combination of orelabrutinib, pomalidomide and rituximab(Pro regimen) in eligible patients, following contrast computed temography(CT) to guide the next treatment. Patients whose lesions have 25% or more reduction will next receive Pro-miniCHOP-like regimen for 6 cycles. Patients with reduction less than 25% will receive R-miniCHOP-like regimen also for 6 cycles. After that, maintenance therapy with pomalidomide for two years will be given to patients undergoing Pro-miniCHOP-like regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically or Cytologically confirmed newly diagnosed untreated DLBCL;
2. There is at least one radiographically measurable lesion (i.e., ≥ 15mm in diameter);
3. Age ≥ 70 years;
4. Life expectancy >3 months;
5. Patients with proper organic function (alanine aminotransferase, bilirubin, creatinine < 3 times the upper limit of normal; cardiac ejection fraction ≥ 50%; SPO2>90% under non-oxygenated conditions).
6. Written informed consent obtained from the subject.

Exclusion Criteria:

1. Patients with severe liver and kidney dysfunction (alanine aminotransferase, bilirubin, creatinine > 3 times the upper limit of normal);
2. Patients with organic heart disease with clinical symptoms or cardiac dysfunction (NYHA grade ≥2);
3. Uncontrolled active infection;
4. Patients with central nervous system DLBCL;
5. A history of vascular embolism;
6. Co-existence of other tumors;
7. Systemic corticosteroid therapy is needed;
8. Any other psychological conditions that prevent patients from participating in the study or signing the informed consent form.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2026-07-03 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) after Pro-miniCHOP-like regimen | At the end of cycle 6 (each cycle is 21 days)
  The rate of patients who achieved complete response and partial response after Pro-miniCHOP-like regimen.
Complete Response Rate(CRR) after Pro-miniCHOP-like regimen | At the end of cycle 6 (each cycle is 21 days)
  The rate of patients who achieved complete response after Pro-miniCHOP-like regimen.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events, treatment-related adverse events and serious adverse events | Initiation of study drug until 28 days after last dose
  The safety and tolerability of the therapeutic regimen measured by the incidence of Treatment-Emergent Adverse Events, Treatment-Related Adverse Events and Serious Adverse Events.
Overall Response Rate(ORR) after Pro induction regimen | At the end of a cycle 1 of induction therapy period (each cycle is 21 days)
  The rate of patients who achieved complete response and partial response after Pro induction regimen.
Complete Response Rate(CRR) after Pro induction regimen | At the end of a cycle 1 of induction therapy period (each cycle is 21 days)
  The rate of patients who achieved complete response after Pro induction regimen.
Overall Survival (OS) | Up to 2 years after the end of last patient's treatment
  OS will be assessed from the first drug given to date of death or end of follow-up.
Progression Free Survival (PFS) | Up to 2 years after the end of last patient's treatment
  PFS will be assessed from the first drug given to date of progression, relapse, death or end of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
All the data would be available at the First Affiliated Hospital and other researchers after the end of the study.
Supporting Information: Study Protocol, SAP
Time Frame: After the end of the study